CLINICAL TRIAL: NCT07367997
Title: Comparative Effectiveness of Verbal Instruction Versus Simulation Video Education Among Cancer Patients Undergoing Radiation Therapy in Lower Middle Income Country Centre: A Randomized Controlled Trial
Brief Title: Comparative Effectiveness of Verbal Instruction Versus Simulation Video Education Among Cancer Patients Undergoing Radiation Therapy
Acronym: CARE-RT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jinnah Postgraduate Medical Centre (Other Government)
Responsible Party: Principal Investigator, Fatima Shaukat, Consultant Radiation Oncologist, Jinnah Postgraduate Medical Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NO.F.2-81/2024-GENL/94/JPMC
Record Dates: First submitted 2026-01-01; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Cancer (Solid Tumors); Cancer and / or Hematological Malignancy
Keywords: Radiation Education
MeSH Terms: conditions — Neoplasms; Hematologic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video Group (Experimental): Patients will receive a WhatsApp message containing the educational video prior to their consultation.
  Interventions: Behavioral: Radiotherapy-Specific Educational Video
- Verbal Instruction Group (No Intervention): Patients will receive a standard verbal education from a radiation oncologist during their consultation.

INTERVENTIONS:
Behavioral: Radiotherapy-Specific Educational Video — This intervention consists of a radiotherapy-specific, physician-led educational video delivered prior to the first radiation oncology consultation. The video was locally developed, filmed within the actual CyberKnife and Tomotherapy facility, and features real radiation oncologists, residents, and departmental staff familiar to patients. It demonstrates real simulation rooms, immobilization devices, and treatment machines that patients will encounter during their care.
  The video is 3.5 minutes in duration, delivered in Urdu, the native language of the study population, and specifically designed for radiation therapy-naïve patients in a lower-middle-income country setting. Content includes an overview of radiation therapy, simulation procedures, treatment delivery, common side effects, and post-treatment follow-up.
  Arms: Video Group

SUMMARY:
The goal of this Randomized Controlled Trial is to compare the effectiveness of radiotherapy-specific, physician-led educational videos introduced before the initial Radiation Therapy consultation .

The primary objective is to assess the impact on patient-reported knowledge of RT, with secondary objectives including assessment of patient-reported anxiety and satisfaction with the educational process.

Patients will be randomly assigned to two groups.

1. Video Group - Patients will receive a WhatsApp message containing the educational video prior to their consultation.
2. Verbal Instruction Group - Patients will receive standard verbal education from a radiation oncologist during their consultation.

The participants will fill Pre and post intervention questionnaire forms

DETAILED DESCRIPTION:
The stress and fatigue associated with cancer treatment are significant concerns that can greatly affect a patient's quality of life. Few studies discussed how common and debilitating cancer-related fatigue can be, highlighting the need for better educational tools to help patients manage their treatment and its side effects. Providing clear, engaging information through videos could help reduce anxiety and make the treatment process less overwhelming for patients.

This study aims to evaluate the effectiveness of radiotherapy-specific, physician-led educational videos introduced before the initial RT consultation. The primary objective is to assess the impact on patient-reported knowledge of RT, with secondary objectives including assessment of patient-reported anxiety and satisfaction with the educational process. Through this approach, we aim to contribute to emerging strategies that optimize patient preparedness and emotional well-being in radiation oncology

Video Development

A single educational video was developed to provide a general overview of radiation therapy for cancer patients undergoing treatment at the Cyber Knife and Tomotherapy Centre, JPMC. The video was designed to enhance patient understanding of the radiation treatment process, and reduce anxiety The volunteers of the student led forum Tumor Board Establishment Facilitation Forum (TEFF), were approached to direct, organize, and film the video. The content of video was developed by a team of radiation oncology from Pakistan and Canada. The video was created in Urdu, the native language of Pakistan, ensuring accessibility for a broad patient population. It was approximately 3.5 minutes long. The editing process was iterative, involving multiple draft scripts and a trial video. Feedback on content, style, and delivery was gathered from all stakeholders before finalizing the videos. The video was assessed using the Patient Education Materials Assessment Tool for Audiovisual Materials (PEMAT-A/V), scoring 100% on understandability and 100% on action ability.

Physicians, resident medical officers, and departmental staff participated in the video, each signing a Consent to Photograph release form. The videos include sections on overview, simulation, treatment, side effects, and post-treatment follow-up.

Study Design This is a Phase 2, single-center, randomized controlled trial (RCT) designed to compare the effectiveness of verbal instruction versus simulation video education among cancer patients undergoing radiation therapy. The study will be conducted at JPMC's Cyber Knife and Tomotherapy Centre, a specialized facility providing cost-free radiation therapy services in Karachi, Pakistan 100 Patients will be randomly assigned to two groups. Randomization will be performed using an online randomization tool (www.randomizer.org) at a 1:1 ratio:

1. Video Group - Patients will receive a WhatsApp message containing the educational video prior to their consultation.
2. Verbal Instruction Group - Patients will receive a standard verbal education from a radiation oncologist during their consultation.

Educational videos specific to our department or physicians are not previously available. Patients scheduled for a simulation, who agree to participate will be sent either to video group or verbal instruction group as per randomization Participants

Patients will be recruited in a span of 6 months. Eligible participants meet the following criteria:

* Diagnosed with cancer and scheduled for radiation therapy at Tomotherapy unit of Cyber knife and Tomotherapy Centre of JPMC.
* Fluent in Urdu.
* No prior experience with radiation therapy.
* Must have smart phone All patients will be offered to participate. Those who did not consent will be excluded.

Outcome Measures

Primary and secondary outcomes will be assessed using validated patient-reported surveys at two time points:

1. Pre-consultation survey - Administered before the radiation oncology consultation to assess baseline patient reported understanding, knowledge and expectations for RT simulation process. It also assesses anxiety and fear related to radiation treatment.
2. Post-consultation survey - Administered after the consultation to measure improvement in understanding, treatment confidence, and satisfaction.

Responses will be collected on a 5-point Likert scale, and comparisons between the two groups will be analyzed to determine the impact of video education versus verbal instruction.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cancer and scheduled for radiation therapy at Tomotherapy unit of Cyber knife and Tomotherapy Centre of JPMC.
* Fluent in Urdu.
* No prior experience with radiation therapy.
* Must have smart phone

Exclusion Criteria:

Patients who either refused consent or were ineligible based on the study's inclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
''Change in Patient-Reported Understanding of Radiation Therapy Between Pre- and Post-Consultation Assessments'' | Baseline and immediately post- educational intervention (same-day assessment)
  The primary outcome of this study is the change in patient-reported knowledge and understanding of radiation therapy (RT) following exposure to educational intervention.
  This outcome is measured by comparing pre- and post-consultation knowledge and understanding scores between the two study arms (video education vs. verbal instruction) using a self-administered 5-point Likert questionnaire (1 = very poor, 5 = excellent). Higher scores indicate better understanding. Anxiety is measured on a 10-point Visual Analog Scale (0 = no anxiety, 10 = maximum), with higher scores indicating worse anxiety.
  The questionnaire evaluates patient understanding across key domains of the radiation therapy process, including RT purpose and goals, simulation and immobilization, treatment delivery, expected side effects, and follow-up. The primary endpoint is the mean change in composite knowledge score from baseline to post-consultation, with greater improvement indicating better understanding.

CONTACTS AND LOCATIONS:
Overall Officials: Fatima Shaukat, MBBS, FCPS, Principal Investigator — Patients Aid Foundation, JPMC; YUMNA AHMED, MBBS, FCPS, Study Director — Patients Aid Foundation, JPMC; Rabia Tahseen, MBBS, FCPS, Study Chair — Patients Aid Foundation, JPMC; Agha Muhammad Hammad Khan, MBBS, FCPS, Study Director — Ziauddin university Hospital